CLINICAL TRIAL: NCT05742438
Title: Effect of Dexmedetomidine Infusion, Lidocaine Infusion, and Intrathecal Morphine Injection on Biomarker for Perioperative Stress and Immune Response, and Cancer Progression and Metastasis in Colorectal Cancer Surgery
Brief Title: Effects of Dexmedetomidine/Lidocaine/Intrathecal Morphine on Cancer Metastasis Biomarker After Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Korea Institute of Science and Technology (Other)
Responsible Party: Principal Investigator, MiHye Park, assistant professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SMC 2022-10-021-002
Record Dates: First submitted 2023-02-06; First posted 2023-02-24 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer; Anesthesia; Cancer Metastatic; Inflammation
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Inflammation | interventions — Lidocaine; Dexmedetomidine; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lidocaine group (Active Comparator): A loading dose of 1.5mg/kg lidocaine will be infused for 10 minutes during anesthesia induction. During the surgery and post-anaesthesia care unit (PACU) stay, 1.5 mg/kg/h of lidocaine were continuously infused until the patient was transferred to the general ward.
  Interventions: Drug: Lidocaine IV
- Dexmedetomidine group (Active Comparator): A loading dose of 0.3mcg/kg dexmedetomidine will be infused for 10 minutes during anesthesia induction. During the surgery and PACU stay, 0.3 mcg/kg/h of dexmedetomidine were continuously infused until the patient was transferred to the general ward.
  Interventions: Drug: Dexmedetomidine IV
- Intrathecal Morphine group (Active Comparator): 200~300mcg of Intrathecal morphine will be injected at the anesthesia induction for colorectal surgery.
  Interventions: Drug: intrathecal morphine

INTERVENTIONS:
Drug: Lidocaine IV — Continuous intravenous infusion of lidocaine
  Other Names: Lidocaine
  Arms: Lidocaine group
Drug: Dexmedetomidine IV — Continuous intravenous infusion of dexmedetomidine
  Other Names: Precedex
  Arms: Dexmedetomidine group
Drug: intrathecal morphine — intrathecal morphine injection
  Other Names: Morphine
  Arms: Intrathecal Morphine group

SUMMARY:
This is a prospective randomized controlled trial. Investigators aimed to compare the effect of three different anesthetic adjuvants (continuous infusion of lidocaine or dexmedetomidine, intrathecal morphine injection) on the biomarker for cancer recurrence and metastasis.

Patients undergoing elective colorectal cancer surgery will be randomly allocated to three parallel arms and the biomarkers for cancer recurrence and metastasis, inflammation, and immune response will be compared. And we will compare the clinical outcomes in the three method.

DETAILED DESCRIPTION:
Perioperative period is critical in determining the risk of postoperative metastatic disease. Surgical damage and related stress response could suppress cell-mediated immunity and facilitate malignant cell survival, motility, invasion and proliferation. Increasing evidence supported that the continuous infusion of lidocaine or dexmedetomidine, or intrathecal morphine were associated with the reduction of postoperative pain and opioid consumption and improved the quality of recovery.

Also, they were reported to decrease perioperative inflammatory responses and preserve immune response which is known to be critical in anti-metastatic process during perioperative period. However, no comparison was conducted among these anesthetic adjuvants. Thus, Investigators try to evaluate the effect on the biomarkers and clinical outcomes in the three methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were scheduled for elective colorectal cancer surgery American Society of Anesthesiologists physical status of I-III

Exclusion Criteria:

* Atrioventricular conduction disorder
* Having Bradycardia (<50 bpm)
* Severe pulmonary dysfunction in pulmonary function test
* High risk for cardiovascular complications(expected postoperative event >5%)
* Allergy or hypersensitivity reaction to each adjuvant.
* History or risk factors for Malignant hyperthermia
* Body mass index >40 kg/m2

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-08-05 (Actual)

PRIMARY OUTCOMES:
MMP-9 | 1 hour after surgery
  plasma Matrix metalloproteinase-9

SECONDARY OUTCOMES:
MMP-9 | at the induction of anesthesia
  plasma Matrix metalloproteinase-9, on the morning of postoperative day 1
MMP-2 | at the inudction of anesthesia, 1 hour after surgery, 1 day after surgery
  plasma Matrix metalloproteinase-2
IL-6 | at the inudction of anesthesia, 1 hour after surgery, 1 day after surgery
  Interleukin-6
VEGF | at the inudction of anesthesia, 1 hour after surgery, 1 day after surgery
  vascular endothelial growth factor
lymphocyte subset | at the inudction of anesthesia, 1 hour after surgery, 1 day after surgery
  CD3+CD4+ (helper T cells), CD3+CD8+ (cytotoxic T cells), CD3-CD16+CD56+ (Natural killer(NK) cells), CD3+CD16+CD56+ NK T cell, CD39+, CD73+, CD39+CD73+ expressions on CD4+ and CD8+ T cells
numeric rating scale | within 3 days after the surgery (1, 6, 24, 48, 72 hour after surgery)
  Pain severity with numeric rating scale for postoperative pain, the value range (0~10), a higher score means more painful
Opioid consumption | within 3 days after the surgery (1, 6, 24, 48, 72 hour after surgery)
  morphine equivalent unit of opioid consumption
postoperative nausea/vomiting | within 3 days after the surgery (1, 6, 24, 48, 72 hour after surgery)
  the requirement of rescue antiemetic
Time to flatus | within 7 days after the surgery
  from the end of surgery to the time of first flatus
Hospital length of stay | Until the discharge (up to postoperative day 30)
  from the end of surgery to patient discharge
respiratory depression | during the night of surgery
  pulse oximetry value < 92% or the need for reintubation.
urinary retention | within 7 days after the surgery
  need for in-and-out catheterization or reinsertion of an indwelling urinary catheter during the hospital stay after the original urinary catheter was removed, and re-operation
Headache and itching sensation | within 3 and 1 day after surgery, respectively
  orthostatic headache and itching sensation
reoperation and readmission rate | within 1 month after surgery and discharge, respectively
  Reoperation was defined as any surgical procedure performed under general or regional anaesthesia for treatment of complications related to the initial operation within 30 days after surgery.
  Readmission was defined as any hospital admission occurring after discharge within 30 days from the index surgery, specifically related to postoperative complications or management associated with the initial surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Mihye Park, MD, PhD, Study Director — Samsung Medical Center
Locations (1):
- Samsung medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levins KJ, Prendeville S, Conlon S, Buggy DJ. The effect of anesthetic technique on micro-opioid receptor expression and immune cell infiltration in breast cancer. J Anesth. 2018 Dec;32(6):792-796. doi: 10.1007/s00540-018-2554-0. Epub 2018 Sep 18. PMID 30229370
- [Background] Wall TP, Buggy DJ. Perioperative Intravenous Lidocaine and Metastatic Cancer Recurrence - A Narrative Review. Front Oncol. 2021 Aug 2;11:688896. doi: 10.3389/fonc.2021.688896. eCollection 2021. PMID 34408981
- [Background] Galos EV, Tat TF, Popa R, Efrimescu CI, Finnerty D, Buggy DJ, Ionescu DC, Mihu CM. Neutrophil extracellular trapping and angiogenesis biomarkers after intravenous or inhalation anaesthesia with or without intravenous lidocaine for breast cancer surgery: a prospective, randomised trial. Br J Anaesth. 2020 Nov;125(5):712-721. doi: 10.1016/j.bja.2020.05.003. Epub 2020 Jun 29. PMID 32616309
- [Background] Wang K, Wu M, Xu J, Wu C, Zhang B, Wang G, Ma D. Effects of dexmedetomidine on perioperative stress, inflammation, and immune function: systematic review and meta-analysis. Br J Anaesth. 2019 Dec;123(6):777-794. doi: 10.1016/j.bja.2019.07.027. Epub 2019 Oct 24. PMID 31668347
- [Background] Liu Y, Sun J, Wu T, Lu X, Du Y, Duan H, Yu W, Su D, Lu J, Tian J. Effects of serum from breast cancer surgery patients receiving perioperative dexmedetomidine on breast cancer cell malignancy: A prospective randomized controlled trial. Cancer Med. 2019 Dec;8(18):7603-7612. doi: 10.1002/cam4.2654. Epub 2019 Oct 30. PMID 31663690
- [Background] Le-Wendling L, Nin O, Capdevila X. Cancer Recurrence and Regional Anesthesia: The Theories, the Data, and the Future in Outcomes. Pain Med. 2016 Apr;17(4):756-75. doi: 10.1111/pme.12893. Epub 2016 Feb 2. PMID 26441010